CLINICAL TRIAL: NCT04461743
Title: Microcirculation Evolution in Patients After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Southeast University, China, Southeast University, China
Other Study IDs: 2020
Record Dates: First submitted 2020-05-31; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Patients After Cardiac Surgery
Keywords: microcirculation; cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with normal lac
  Interventions: Other: No intervention
- Patients with abnormal lac
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, regular therapy

SUMMARY:
We evaluated the impact on macrocirculatory hemodynamics and microcirculation in patients after cardiac surgery and compared the evolutions of those parameters between patients with tissue hypoperfusion and normal perfusion. Consecutive patients after cardiac surgery who required mechanical ventilation and for whom sublingual microcirculation measurements were possible enrolled.

DETAILED DESCRIPTION:
We evaluated the impact on macrocirculatory hemodynamics and microcirculation in patients after cardiac surgery and compared the evolutions of those parameters between patients with tissue hypoperfusion and normal perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients after cardiac surgery.
* Patients whom sublingual microcirculation measurements were possible.

Exclusion Criteria:

* moribund patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients after cardiac surgery who required mechanical ventilation and for whom sublingual microcirculation measurements were possible.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Microcirculation | Extubation
  PPV and MFI

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, Principal Investigator — Southeast University
Locations (1):
- Department of Critical Care Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided